CLINICAL TRIAL: NCT05017701
Title: Feasibility of Bridge for Post-Operative Pain Management in Hip Arthroplasty
Status: Terminated | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CHEL0001
Record Dates: First submitted 2021-07-30; First posted 2021-08-24 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Unapproved Device: Yes

ARMS (2):
- Bridge device (Experimental): The active Bridge device delivers electrical stimulation to the cranial and occipital nerves.
  Interventions: Device: Bridge device
- Sham device (Sham Comparator): The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Bridge device — Bridge is a percutaneous nerve field stimulation device which uses alternating currents of stimulation over a large field and with higher voltage in order to influence central pain areas.
  Arms: Bridge device
Device: Sham device — The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses.
  Arms: Sham device

SUMMARY:
The aim of this research study is to gather data regarding the feasibility of the Bridge system for the management of pain following total hip arthroplasty (THA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject scheduled for elective primary unilateral total hip arthroplasty (THA)
* Subject opioid use is less than 60 milligram morphine equivalent for the last 30 days
* Subject has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects who are pregnant or breastfeeding
* Subjects with cardiac pacemakers or other implanted devices (e.g. vagal nerve simulators), hemophilia or psoriasis vulgaris
* Subjects with a history of active depression, anxiety or catastrophizing
* Subjects with active alcoholism or drug abuse
* Subjects with severe chronic pain condition that requires daily preoperative opioid dependence
* Subjects deemed not suitable for the study at the discretion of the principal investigator
* Subjects who are concurrently participating in any other research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bridge Device | Sham Device
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bridge Device | Sham Device | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Opioid Consumption Between Active and Sham Arms.
Description: The sample size is well below the threshold needed to reliably assess outcomes and perform statistical comparisons. As a result, we have provided the raw data for comparison of opioid consumption between the two groups.
Time Frame: Day of surgery to Day 5 (120 hours) post-op
Population: The study was terminated prematurely due to sponsor decision, with no clinical rationale for the termination. This was a feasibility study and the test device was deemed "end-of-life" by the manufacturer. Only 5 subjects were enrolled out of the 60 anticipated -2 with active devices and 3 with sham devices. All available demographic and outcome measure data from the limited sample size have been reported. Further data reporting would be statistically inappropriate due to the sample size.
Measure: Number; unit: doses
Arm/Group | Bridge Device | Sham Device
Number analyzed (Participants) | 2 | 3
doses
  Oxycodone 5mg | 1 | 33
  Tramadol 50mg | 0 | 5
  Meloxicam 15mg | 0 | 7

2. Secondary Outcome: Change in Pain Between Active and Sham Arms as Measured Using the Numeric Rating Scale.
Description: Pain scores using a numerical scale will be collected at rest and movement and will be obtained prior to surgery, in the recovery room, prior to leaving the recovery room, every 6 hours during the first 24 hrs, and at 48, 72, 96 and 120 hours post-operatively. Subjects will use a 0-10 numeric scale (0 indicating no pain and 10 indicating extreme pain).
Time Frame: Day of surgery to Day 5 (120 hours) post-op
Population: The study was terminated prematurely due to sponsor decision, with no clinical rationale for the termination. This was a feasibility study and the test device was deemed "end-of-life" by the manufacturer. Only 5 subjects were enrolled out of the 60 anticipated -2 with active devices and 3 with sham devices. All available demographic and outcome measure data from the limited sample have been reported. Further data reporting would be statistically inappropriate due to the sample size.
Measure: Number; unit: score on a scale
Groups:
- Subject 1 - Bridge Device; Subject 2 - Bridge Device: The active Bridge device delivers electrical stimulation to the cranial and occipital nerves.
  Bridge device: Bridge is a percutaneous nerve field stimulation device which uses alternating currents of stimulation over a large field and with higher voltage in order to influence central pain areas.
- Subject 3 - Sham Device; Subject 4 - Sham Device; Subject 5 - Sham Device: The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses
  Sham device: The sham device has the same appearance and will require the same placement technique as the Bridge (active) device but will not deliver electrical impulses.
Arm/Group | Subject 1 - Bridge Device | Subject 2 - Bridge Device | Subject 3 - Sham Device | Subject 4 - Sham Device | Subject 5 - Sham Device
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
score on a scale
  6 hours post-op | 9 | 1 | 7 | 5 | 5
  12 hours post-op | 7 | 1 | 7 | 4 | 8
  18 hours post-op | 7 | 2 | 7 | 2 | 6
  Day 1 (24 hours) post-op | 8 | 0 | 6 | 1 | 6
  Day 2 (48 hours) post-op | 4 | 1 | 4 | 4 | 5
  Day 3 (72 hours) post-op | 4 | 1 | 5 | 3 | 4
  Day 4 (96 hours) post-op | 3 | 4 | 5 | 2 | 3
  Day 5 (120 hours) post-op | 4 | 1 | 3 | 3 | 3

3. Secondary Outcome: Change in Postoperative Nausea Between Active and Sham Arms as Measured Using a Postoperative Nausea and Vomiting Rating Scale.
Description: Postoperative nausea and vomiting will be evaluated from immediately after surgery through postoperative day 5, using a 0-10 scale (0 indicating no nausea and 10 indicating extreme nausea).
Time Frame: Day of surgery to Day 5 (120 hours) post-op
Population: as for outcome 2
Measure: Number; unit: score on a scale
Arm/Group | Subject 1 - Bridge Device | Subject 2 - Bridge Device | Subject 3 - Sham Device | Subject 4 - Sham Device | Subject 5 - Sham Device
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
score on a scale
  6 hours post-op | 0 | 0 | 0 | 0 | 0
  12 hours post-op | 0 | 0 | 0 | 0 | 0
  18 hours post-op | 0 | 0 | 0 | 0 | 0
  Day 1 (24 hours) post-op | 0 | 0 | 3 | 0 | 0
  Day 2 (48 hours) post-op | 0 | 0 | 0 | 0 | 0
  Day 3 (72 hours) post-op | 0 | 0 | 0 | 0 | 0
  Day 4 (96 hours) post-op | 0 | 0 | 0 | 0 | 0
  Day 5 (120 hours) post-op | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Functional Recovery Between Active and Sham Arms Assessed Using the Timed Up and Go (TUG) Assessment Collected on Post-Op Day 30
Description: Functional recovery will be assessed daily from day of surgery to post-op day 5, using the Timed Up and Go assessment to assess mobility.
Time Frame: Day of surgery to post-operative day 30.
Population: No data was collected for this outcome measure. The study was terminated prematurely due to sponsor decision, with no clinical rationale for the termination. This was a feasibility study and the test device was deemed "end-of-life" by the manufacturer. Only 5 subjects were enrolled out of the 60 anticipated -2 with active devices and 3 with sham devices. All available demographic and outcome measure data from the limited sample have been reported.
Arm/Group | Bridge Device | Sham Device
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Functional Recovery Between Active and Sham Arms Assessed Using the 12-Item Short Form Survey (SF-12) Collected on Post-Op Day 30
Description: Subjects will also complete the 12-Item Short Form Survey (SF-12) on Post-Op day 30 to evaluate quality of recovery.
Time Frame: Day of surgery to post-operative day 30.
Population: as for outcome 4
Arm/Group | Bridge Device | Sham Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of surgery to post-operative day 5
Arm/Group | Bridge Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT05017701/Prot_SAP_000.pdf